CLINICAL TRIAL: NCT06655376
Title: Delayed ARIES: Aspirin and Hemocompatibility Events in Advanced Heart Failure Patients Chronically Supported with a Left Ventricular Assist Device
Brief Title: Aspirin and Hemocompatibility Events in Chronic Advanced Heart Failure Patients with Assist Device
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Weill Medical College of Cornell University (Other)
Responsible Party: Principal Investigator, Nir Uriel, Professor of Cardiology (in Medicine), Columbia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AAAV3358
Record Dates: First submitted 2024-10-22; First posted 2024-10-23 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-10

CONDITIONS: Bleeding; Clot Blood
MeSH Terms: conditions — Hemorrhage; Thrombosis | interventions — Aspirin; Warfarin; acarboxyprothrombin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Warfarin without Aspirin (Experimental): Participants will only take Warfarin.
  Interventions: Drug: Warfarin
- Warfarin and Aspirin (Active Comparator): This is the control arm. Participants will take Warfarin and aspirin, which is the standard of care.
  Interventions: Drug: Aspirin; Drug: Warfarin

INTERVENTIONS:
Drug: Aspirin — 81-100 mg, oral
  Other Names: ASPIRIN® tablets
  Arms: Warfarin and Aspirin
Drug: Warfarin — Warfarin dose will be adjusted per patient for a goal INR 2-3. The individualized daily dose could range anywhere from 0.5-2 mg to 5-7 mg. Oral.
  Other Names: Vitamin K antagonist; COUMADIN

SUMMARY:
Heart failure is a world epidemic. LVADs are increasingly used as they have demonstrated improved survival rates compared to optimal medical management. Improving outcomes have been seen with the newer LVAD technology, the HeartMate 3 (Abbott, Chicago, IL), however, hemocompatibility related adverse events, including thrombosis and bleeding, are still a major cause of morbidity and mortality. The recent ARIES trial showed that in patients with advanced heart failure treated with a HeartMate3 LVAD, avoidance of aspirin as part of an antithrombotic regimen, which includes vitamin K antagonist (VKA), is not inferior to a regimen containing aspirin, does not increase thromboembolism risk, and is associated with a reduction in bleeding events.

This clinical investigation is a prospective, randomized, controlled study of advanced heart failure patients supports with the HeartMate3 for more then 3 months with two different antithrombotic regimens: VKA with and without aspirin. The objective of this investigation is to study the safety and efficacy of an antithrombotic regimen without antiplatelet therapy.

DETAILED DESCRIPTION:
Objective: To study the safety and efficacy of an anti-platelet-free antithrombotic regimen in patients with advanced heart failure who are chronically supported with the HeartMate 3 LVAD.

Hypothesis: The withdrawal of aspirin from the antithrombotic regimen of HeartMate3 LVAD patients will not adversely affect safety and efficacy and may reduce non-surgical bleeding.

Clinical Investigation Design: This is a prospective, randomized, controlled clinical investigation of advanced heart failure patients who are chronically supported with the HeartMate 3 LVAD. The study will compare two different antithrombotic regimens: VKA with aspirin versus VKA without aspirin.

End points:

Primary end point:

* Composite of Survival free of any major hemocompatibility related adverse event at 1-year post randomization.

  1. Major Hemocompatibility Related Adverse Event: Stroke, Pump Thrombosis (suspected or confirmed), major non surgical Bleeding (moderate or severe) (including intracranial bleeds that do not meet the stroke definition), Arterial Peripheral Thromboembolism

     Secondary end point:
* Non-surgical Major Hemorrhagic Events
* Non-surgical Major Thrombotic Events
* Survival
* Stroke Rates
* Pump Thrombosis Rates
* Bleeding Rates, including:

  * Non-surgical Bleeding
  * Moderate Bleeding
  * Severe Bleeding
  * Fatal Bleeding
  * GI Bleeding Descriptive endpoints
* Hemocompatibility score:

a tiered hierarchal score that weighs each hemocompatibility related adverse event by its escalating clinical relevance⁸

* Rehospitalizations
* Economic Cost Implications
* Subgroup analysis (patients with increased bleeding/thrombotic risk (i.e prior HRAE events)

Number of Subjects Required for Inclusion in Clinical Investigation:

Based on ARIES results, 58 patients will need to be enrolled in each arm (116 total) to achieve 80% power to prove that the non-aspirin group is non-inferior to the aspirin group using a non-inferiority margin of 15% with the Farrington-Manning risk difference approach to non-inferiority at a one-sided alpha = 0.05. To account for an expected 10% dropout rate, up to 128 patients will be randomized in the trial.

ELIGIBILITY:
Inclusion Criteria:

* Participant will have HeartMate3 LVAD implanted > 3 months before enrollment.
* >18 years old
* Treated with aspirin and VKA
* Participant must provide written informed consent prior to any clinical investigation-related procedure

Exclusion Criteria:

* Investigator-mandated antiplatelet therapy for other conditions (including mandated presence or absence of antiplatelet agent)
* Participation in any other clinical investigation(s) involving an MCS device, or interventional investigation(s) likely to confound study results or affect study outcome
* Presence of other anatomic or comorbid conditions, or other medical, social, or psychological conditions that, in the investigator's opinion, could limit the subject's ability to participate in the clinical investigation or to comply with follow-up requirements, or impact the scientific soundness of the clinical investigation results
* Pregnant and on appropriate contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2024-10-02 (Actual); Primary Completion 2027-04-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Number of survival free patients of any major hemocompatibility related adverse events. | 1 year post implant
  A Major Hemocompatibility Related Adverse Event is defined as: Stroke, Pump Thrombosis (suspected or confirmed), major non-surgical Bleeding (moderate or severe) (including intracranial bleeds that do not meet the stroke definition), Arterial Peripheral Thromboembolism. The events will be recorded and tallied per patient.

SECONDARY OUTCOMES:
Number of Non-surgical Major Hemorrhagic Events | 1 year
  The following types of events will be recorded and tallied. MODERATE or severe bleeding as defined in the protocol. SEVERE or overt bleeding plus hemoglobin drop of 3 to < 5 g/dL (provided hemoglobin drop is related to bleed).
  Any transfusion with overt bleeding. Cardiac tamponade. Bleeding requiring surgical intervention for control (excluding dental, nasal, skin, or hemorrhoid).
  Hypotension attributable to bleeding.
Number of Non-surgical Major Thrombotic Events | 1 year
  The following types of events will be recorded and tallied:
  The Device Thrombosis, Stroke, Arterial non-CNS thromboembolism.
Survival Rate | 1 year
  Patients who survive at 1 year post implant will be recorded and tallied.
Stroke Incidence | 1 year
  The following types of events will be recorded and tallied. Ischemic Stroke Hemorrhagic Stroke
Pump Thrombosis Incidence | 1 year
  pump thrombosis or suspected will be recorded and tallied.
Bleeding Incidence | 1 year
  Bleeding Rates, including Non-surgical Bleeding, Moderate Bleeding, Severe Bleeding, Fatal Bleeding, GI Bleeding will be recorded and tallied.

OTHER OUTCOMES:
Hemocompatibility Score | 1 year
  A tiered hierarchal score that weighs each hemocompatibility related adverse event by its escalating clinical relevance will be recorded and scored.
Number of Rehospitalizations | 1 year
  number of all hospitalizations at 1 year, including number of HF related hospitalizations, will be tallied.
Averaged Days of hospitalization | 1 year
  This is to measure economic cost. Health resource utilization will be assessed by comparing days hospitalized (categorized by intensive care vs general ward) between groups.
Number of patients with increased bleeding/thrombotic risk | 1 year
  Patients with increased events when compared to prior HRAE events will be assessed and tallied.

CONTACTS AND LOCATIONS:
Overall Officials: Nir Uriel, MD, Principal Investigator — Seymour, Paul, and Gloria Milstein Professor of Cardiology at Columbia University
Locations (1):
- Columbia Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided